CLINICAL TRIAL: NCT01712945
Title: Keratinocyte Growth Factor - Promoting Thymic Reconstitution and Preventing Autoimmunity After Alemtuzumab (Campath-1H) Treatment of Multiple Sclerosis
Brief Title: Keratinocyte Growth Factor to Prevent Autoimmunity After Alemtuzumab Treatment of Multiple Sclerosis
Acronym: CAM-THY
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: interim anlaysis failed: palifermin does not promote thymopoeisis after alemtuzumab
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Alasdair Coles, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EudraCT 2011-005606-30
Record Dates: First submitted 2012-10-19; First posted 2012-10-24 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: Alemtuzumab; Palifermin; Reconstitution; Thymus
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fibroblast Growth Factor 7; Alemtuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palifermin (and Alemtuzumab) (Experimental): Palifermin (Kepivance®), at the maximum identified tolerated dose will be administered by intravenous bolus on days -5, -4. -3 prior to, and on days 8, 9 and 10 after each cycle of alemtuzumab, then again on 3 consecutive days at month 1 and month 3 after each cycle of alemtuzumab. Patients will be observed for adverse reactions for at least 1 to 2 hours following each bolus dose. Initial treatment alemtuzumab will be administered as a fixed total dose of 60 mg IV over 5 consecutive days (12mg/day). For re-treatment at Month 12, alemtuzumab will be administered as a fixed total dose of 36mg IV over 3 consecutive days (12mg/day).
  Interventions: Drug: Palifermin; Drug: Alemtuzumab
- Placebo (and Alemtuzumab) (Placebo Comparator): Initial treatment alemtuzumab will be administered as a fixed total dose of 60 mg IV over 5 consecutive days (12mg/day). For re-treatment at Month 12, alemtuzumab will be administered as a fixed total dose of 36mg IV over 3 consecutive days (12mg/day).
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Palifermin — Palifermin (Kepivance®) administered by intravenous bolus on days -5, -4. -3 prior to, and on days 8, 9 and 10 after each cycle of alemtuzumab, then again on 3 consecutive days at month 1 and month 3 after each cycle of alemtuzumab. Patients will be observed for adverse reactions for at least 1 to 2 hours following each bolus dose.
  Other Names: Kepivance; keratinocyte growth factor
  Arms: Palifermin (and Alemtuzumab)
Drug: Alemtuzumab — Initial treatment alemtuzumab will be administered as a fixed total dose of 60 mg IV over 5 consecutive days (12mg/day). For re-treatment at Month 12, alemtuzumab will be administered as a fixed total dose of 36mg IV over 3 consecutive days (12mg/day).
  Other Names: Campath-1H

SUMMARY:
The purpose of this study is to test a novel strategy to prevent the clinical problem of secondary autoimmunity following alemtuzumab treatment of multiple sclerosis.

The hypothesis is that autoimmunity after alemtuzumab can be prevented by giving a drug that promotes thymic T cell regeneration (Palifermin, Kepivance®).

DETAILED DESCRIPTION:
This is a single-centre, double-blinded, randomised controlled trial of palifermin (Kepivance) vs. placebo in the prevention of autoimmunity following alemtuzumab treatment of multiple sclerosis.

The dose of palifermin (kepivance)used in this trial will be informed by a dose-escalation study.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients
* > 18 years of age, and <50 years of age inclusive
* Diagnosis of MS using McDonald's 2010 criteria, including MRI abnormalities consistent with McDonald's 2010 criteria.
* Onset of first MS symptoms within 10 years on the date the ICF is signed
* EDSS score 0.0 to 5.0 (inclusive) at screening
* At least 2 clinical episodes of MS in the 2 years prior to study entry, with at least 1 attack within 12 months, which may have occurred whilst on disease-modifying therapy, namely any beta interferon or glatiramer acetate.
* Serum IL-7≤7pg/mL

Exclusion Criteria:

* Any progressive form of multiple sclerosis
* Previous thymectomy
* Previous treatment with alemtuzumab, natalizumab, mitoxantrone, cyclophosphomide, cladribine, rituximab or any other immunosuppressant or cytotoxic therapy (other than steroids and disease-modifying therapies listed above)
* History of malignancy
* Personal history of clinically significant autoimmune disease, other than multiple sclerosis (including but not limited to: thyroid disease, immune cytopenias, inflammatory bowel disease, diabetes, lupus, severe asthma)
* Intolerance of pulsed corticosteroids, especially a history of steroid psychosis
* Major systemic disease or other illness that would, in the opinion of the investigator, compromise patient safety or interfere with the interpretation of study results.
* Seropositivity for human immunodeficiency virus (HIV)
* Past or present hepatitis B infection (positive hepatitis B serology)
* Pregnant women or male and female patients who do not agree to use effective contraception during the study.
* Medical, psychiatric, cognitive or other conditions that, in the investigator's opinion, compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study.

Ages: 18 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
incidence of clinical autoimmunity | within 30 months of starting treatment with alemtuzumab
  The primary endpoint is incidence of clinical autoimmunity within 30 months of starting treatment with alemtuzumab

SECONDARY OUTCOMES:
Absolute numbers of naive T cells | within 30 months of starting treatment with alemtuzumab
  Absolute numbers of naive T cells
Safety events | within 30 months of starting treatment with alemtuzumab
  Safety outcomes - incidence and nature of adverse events

OTHER OUTCOMES:
Time at which autoimmunity develops | Within 30 months after alemtuzumab
Reconstitution of lymphocyte subsets | within 30 months of starting treatment with alemtuzumab
  Percentage of naive, central memory, effector memory and effector memory RA cells within the CD4 and CD8 T cell populations
T cell receptor (TCR) clonality | within 30 months of starting treatment with alemtuzumab
  T cell receptor (TCR) clonality
Thymic function | within 30 months of starting treatment with alemtuzumab
  Thymic function - determined by measuring TRECs
Thymic volume | within 30 months of starting treatment with alemtuzumab
  Thymic volume and density - as assessed by non-contrast enhanced, low dose CT scans of the chest performed at baseline and month 6.
Thymic density | within 30 months of starting treatment with alemtuzumab
  Thymic volume and density - as assessed by non-contrast enhanced, low dose CT scans of the chest performed at baseline and month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Coles, Phd FRCP, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Coles AJ, Fox E, Vladic A, Gazda SK, Brinar V, Selmaj KW, Bass AD, Wynn DR, Margolin DH, Lake SL, Moran S, Palmer J, Smith MS, Compston DA. Alemtuzumab versus interferon beta-1a in early relapsing-remitting multiple sclerosis: post-hoc and subset analyses of clinical efficacy outcomes. Lancet Neurol. 2011 Apr;10(4):338-48. doi: 10.1016/S1474-4422(11)70020-5. PMID 21397567
- [Background] Jones JL, Phuah CL, Cox AL, Thompson SA, Ban M, Shawcross J, Walton A, Sawcer SJ, Compston A, Coles AJ. IL-21 drives secondary autoimmunity in patients with multiple sclerosis, following therapeutic lymphocyte depletion with alemtuzumab (Campath-1H). J Clin Invest. 2009 Jul;119(7):2052-61. doi: 10.1172/JCI37878. Epub 2009 Jun 22. PMID 19546505
- [Background] Cox AL, Thompson SA, Jones JL, Robertson VH, Hale G, Waldmann H, Compston DA, Coles AJ. Lymphocyte homeostasis following therapeutic lymphocyte depletion in multiple sclerosis. Eur J Immunol. 2005 Nov;35(11):3332-42. doi: 10.1002/eji.200535075. PMID 16231285
- [Background] CAMMS223 Trial Investigators; Coles AJ, Compston DA, Selmaj KW, Lake SL, Moran S, Margolin DH, Norris K, Tandon PK. Alemtuzumab vs. interferon beta-1a in early multiple sclerosis. N Engl J Med. 2008 Oct 23;359(17):1786-801. doi: 10.1056/NEJMoa0802670. PMID 18946064
- [Background] Bruinsma M, van Soest PL, Leenen PJ, Lambrecht BN, Cupedo T, Lowenberg B, Cornelissen JJ, Braakman E. Keratinocyte growth factor induces expansion of murine peripheral CD4+Foxp3+ regulatory T cells and increases their thymic output. J Immunol. 2007 Dec 1;179(11):7424-30. doi: 10.4049/jimmunol.179.11.7424. PMID 18025186
- [Background] Miller RD, Caulfield MJ, Calkins CE. Expression and regulation of a recurrent anti-erythrocyte autoantibody idiotype in spleen cells from neonatal and adult BALB/c mice. J Immunol. 1992 Apr 15;148(8):2452-5. PMID 1560201
- [Background] Min D, Panoskaltsis-Mortari A, Kuro-O M, Hollander GA, Blazar BR, Weinberg KI. Sustained thymopoiesis and improvement in functional immunity induced by exogenous KGF administration in murine models of aging. Blood. 2007 Mar 15;109(6):2529-37. doi: 10.1182/blood-2006-08-043794. Epub 2006 Nov 30. PMID 17138819
- [Derived] Coles AJ, Azzopardi L, Kousin-Ezewu O, Mullay HK, Thompson SA, Jarvis L, Davies J, Howlett S, Rainbow D, Babar J, Sadler TJ, Brown JWL, Needham E, May K, Georgieva ZG, Handel AE, Maio S, Deadman M, Rota I, Hollander G, Dawson S, Jayne D, Seggewiss-Bernhardt R, Douek DC, Isaacs JD, Jones JL. Keratinocyte growth factor impairs human thymic recovery from lymphopenia. JCI Insight. 2019 May 7;5(12):e125377. doi: 10.1172/jci.insight.125377. PMID 31063156
- See also: Information for patients on protocol — http://www.colescambridge.org.uk/trial%20participation.htm